CLINICAL TRIAL: NCT02064920
Title: A Clinical Trial to Assess Cognitive Function by Repeated Computerized Testing in Patients With Mild Alzheimer's Disease Treated With Donepezil
Brief Title: Computerized Cognition Testing in Participants With Mild Alzheimer's Disease (AD) Treated With Donepezil (MK-0000-318)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 0000-318
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo for donepezil hydrochloride capsule administered orally once a day for 16 weeks.
  Interventions: Drug: Placebo
- Donepezil (Experimental): During the first 4 weeks, participants received placebo for donepezil. Over the following 2 weeks, participants were treated with donepezil at 5 mg per day. Then, over the remaining 10 weeks were titrated to up to 10 mg per day donepezil based on tolerability.
  Interventions: Drug: Placebo; Drug: Donepezil

INTERVENTIONS:
Drug: Placebo — Placebo for donepezil hydrochloride capsule
Drug: Donepezil — 5 mg donepezil hydrochloride capsule.
  Other Names: Aricept
  Arms: Donepezil
Drug: Donepezil — 10 mg donepezil hydrochloride capsule.
  Other Names: Aricept
  Arms: Donepezil

SUMMARY:
This study aims to determine whether the Cogstate testing battery can detect improvements in cognitive function in participants with mild AD. The primary hypothesis is that for one of the Cogstate battery tests, One Card Learning (OCL), the standard deviation associated with the change from baseline in OCL measurements after 12 weeks of donepezil and placebo treatments is =<0.1

ELIGIBILITY:
Inclusion Criteria:

* Meets listed criteria for a diagnosis of probable AD
* Has a clearly documented history either in medical records or from an informant of cognitive decline over at least 6 months
* Has a reliable partner/caregiver who is willing to provide input by participating in assessments
* Has results of a physical examination and clinical laboratory tests within normal or clinically acceptable limits
* Can communicate with trial staff acceptably, possesses the ability to respond verbally to questions, follow instructions, complete questionnaires, and adhere to visit schedules
* Can read at a 9th grade level or equivalent, and has an acceptable history of academic achievement and/or employment
* Has a magnetic resonance imaging (MRI) scan that rules out non-AD conditions contributing to cognitive dysfunction
* Capably performs the CogState screening battery
* Has adequate visual acuity and function
* Females are not of childbearing potential

Exclusion Criteria:

* Has ever received acetylcholinesterase inhibitors, memantine, or other symptomatic AD treatment including approved medical foods
* Has an uncontrolled, clinically significant medical condition or situation within 3 months prior to screening
* Has had major surgery within 3 months prior to screening
* Has tested positive for human immunodeficiency virus (HIV) or has evidence of an active hepatitis B infection
* Has a history of malignancy within the prior 5 years
* Is unwilling or ineligible to undergo an MRI scan
* Has a history of clinically important structural changes on screening MRI scan
* Has a clinically important history of stroke or a diagnosis of vascular dementia
* Has evidence of a clinically relevant non-AD neurological disorder
* Has a history of head trauma, or serious infectious disease affecting the brain within the prior 3-5 years
* Has evidence of a clinically relevant or unstable psychiatric disorder, excepting major depression in remission
* Has evidence of a current episode of major depression
* Has evidence of Type 4 or Type 5 Suicidal Ideation
* Has clinically significant vitamin B12 or folate deficiency in the 6 months prior to screening
* Is pregnant, attempting to become pregnant or is nursing children
* Has used any investigational drug or participated in any other clinical trial within the prior 30 days
* Has a history of alcoholism or drug dependency/abuse within the last 5 years
* Has a relative contraindication to donepezil including sick sinus syndrome, third degree heart block, active gastrointestinal (GI) bleeding, Zollinger-Ellison syndrome, uncontrolled peptic ulcer disease, or uncontrolled asthma

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04-22 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males and females with mild Alzheimer's Disease (AD) between the ages of 55 and 85 years (inclusive) were enrolled in this trial.
Period: Overall Study
Arm/Group | Placebo | Donepezil
Started | 6 | 30
Treated | 6 | 28 (Two participants discontinued from study prior to treatment)
Completed | 5 | 21
Not Completed | 1 | 9
Not completed — Adverse Event | 0 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Technical Problems | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Donepezil | Total
Number analyzed (Participants) | 6 | 30 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.7 (8.6) | 72.7 (8.7) | 73.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 15 | 17
  Male | 4 | 15 | 19

OUTCOME MEASURES:

1. Primary Outcome: One-card Learning (OCL) Measurement Over 12 Weeks of Treatment
Description: OCL is one of the Cogstate battery of tests, and is a continuous visual recognition task that assesses visual recognition, memory and attention using a pattern separation algorithm. OCL is a score defined as the arcsine transformation of the square root of the proportion of correct responses to 80 OCL questions. The score ranges from 0 to 1.5708 where a higher score means better performance.
Time Frame: Weeks 4, 8, 12 and 16
Population: All participants who received study medication and yielded at least one measurement for that endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Donepezil
Number analyzed (Participants) | 5 | 28
Score on a scale
  Week 4 (n = 5, 28) | 0.954 (0.091) | 0.942 (0.112)
  Week 8 (n = 5, 22) | 0.822 (0.179) | 0.969 (0.104)
  Week 12 (n = 5, 21) | 0.849 (0.132) | 0.984 (0.118)
  Week 16 (n = 5, 21) | 0.961 (0.123) | 0.993 (0.112)
Statistical Analysis 1: Comparison: Placebo vs Donepezil; Change from Week 4 to Week 16 in Standard Deviation (SD) of OCL for Placebo + Donezepil treatment groups combined; Test type: Superiority or Other; Change in SD from Week 4 to Week 16 = 0.005, 95% CI 2-sided [-0.031 to 0.039] — SD of average OCL repeated measurements after 12 weeks of treatment for Placebo + Donezepil treatment groups combined is hypothesized to be ≤ 0.1

2. Secondary Outcome: Percentage of Correct Responses in the OCL Task Over 12 Weeks of Treatment
Description: OCL is one of the Cogstate battery of tests, and is a continuous visual recognition task that assesses visual recognition, memory and attention using a pattern separation algorithm. The percentage of correct responses to 80 OCL questions is defined as the number of correct responses x 100 divided by the number of total responses; and ranges from 0 to 100, where 100 is best, and 0 is the worst outcome.
Time Frame: Weeks 4, 8, 12 and 16
Population: All participants who received study medication and yielded at least one measurement for that endpoint.
Measure: Mean (Standard Deviation); unit: Percentage of Corrrect Responses
Arm/Group | Placebo | Donepezil
Number analyzed (Participants) | 5 | 28
Percentage of Corrrect Responses
  Week 4 (n = 5, 28) | 66.2 (8.3) | 64.9 (10.3)
  Week 8 (n = 5, 22) | 53.7 (17.1) | 67.4 (9.5)
  Week 12 (n = 5, 21) | 56.1 (12.7) | 68.6 (10.4)
  Week 16 (n = 5, 21) | 66.7 (11.6) | 69.5 (9.8)

ADVERSE EVENTS:
Time Frame: Up to Week 18 (approximately up to 129 days)
Description: All participants who received study medication.
Arm/Group | Placebo | Donepezil
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/28
Other Adverse Events (participants affected / at risk) | 3/6 | 9/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Donepezil (N=28)
Chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Donepezil (N=28)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.